CLINICAL TRIAL: NCT03480282
Title: Discussing Stopping Cancer Screening and Prognosis With Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mara Schonberg, Principle Investigator - Staff Physician, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016P000244; R21CA212386 (NIH)
Record Dates: First submitted 2018-03-09; First posted 2018-03-29 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Cancer Screening
Keywords: Life expectancy; Older adults; Primary care; Cancer screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prognosis Information and Provider Scripts (Experimental): Investigators will send the PCP via secure email the patient's prognosis calculated by the Lee-Schonberg index three days before the patient visit. Investigators will also send PCPs information on patient life expectancy from Cho et al.'s US life tables and scripts developed to sensitively include information on patient prognosis when recommending patients stop being screened for cancer. After five of their patients have participated or recruitment goals are met, investigators will ask PCPs to complete a 10 minute web-based questionnaire about their experience.
  Interventions: Other: Prognosis information and Provider Scripts

INTERVENTIONS:
Other: Prognosis information and Provider Scripts — An individualized report including each patient's prognosis will be calculated by the Lee-Schonberg and will include information on patient life expectancy from Cho et al.'s US life tables. This report will be sent to the PCP three days before the patient visit. Example scripts for PCPs to use with patients when discussing life expectancy and stopping cancer screening will be sent with the patient prognostic information.

SUMMARY:
Guidelines recommend not screening adults with <10-year life expectancy for cancer; however, primary care physicians feel uncomfortable talking to older adults about prognosis. The investigators aim to determine whether providing PCPs with scripts on patient prognosis and older adults with information on their prognosis would be useful when recommending stopping cancer screening.

DETAILED DESCRIPTION:
The American Cancer Society and the American Board of Internal Medicine Choosing Wisely Campaign recommend clinicians not screen older adults who have <10 year life expectancy for breast (specific to women) or colorectal cancer (CRC). This is because these patients have little chance of experiencing the life prolonging benefits of cancer screening and instead may only experience harm from being screened. The most concerning harm of cancer screening is overdiagnosis - the diagnosis and treatment of cancers that otherwise would not have caused problems in an older adult's lifetime. Despite this, around half of adults >75 years with <10 year life expectancy are regularly screened for cancer. One reason for the overuse of these tests is that PCPs feel uncomfortable discussing stopping screening with older adults since it requires estimating and discussing patient prognosis. Some PCPs admit to recommending cancer screening to older adults with short life expectancy simply to avoid talking to patients about prognosis. However, by avoiding these discussions, PCPs may be impeding older adults' ability to make informed decisions about their care and may be putting patients at risk of the harms of cancer screening without any chance of benefit. Therefore, the investigators aim to interview PCPs and older adults about their thoughts and feelings on how PCPs may discuss older adults' prognosis in the context of talking about stopping cancer screening. Based on those findings, the investigators will develop strategies for PCPs to use to approach these discussions and will draft scripts to suggest language for PCPs to use when communicating about prognosis when recommending stopping cancer screening. Then, the investigators will study if providing PCPs with these scripts and information about their patients' prognosis is useful. Specifically, the investigators will provide 45 PCPs with information about their patients' prognosis and the example scripts before a clinic visit for up to 5 of their patients. The investigators aim to recruit 90 patients with approximately 5-10 year life expectancy. The investigators will interview PCPs and older adults after these visits to learn how and/or if the prognostic information and the scripts were used. These data are essential for improving the quality of PCP discussions around stopping cancer screening and will ultimately improve the care of older adults.

Specific Aims:

1. To learn from PCPs and older adults about how to discuss patient prognosis when recommending stopping cancer screening and to develop strategies for having these discussions.
2. To study whether providing information on patient prognosis and scripts for discussing patient prognosis when recommending stopping cancer screening are useful to PCPs and older adults.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Aged 76 to 89 years
* Scheduled for a routine visit or physical with their PCP in the next 3-12 weeks
* Patient aged 76-79 must have a least one Charlson Comorbidity
* Patient must have undergone CRC screening within the last 10 years
* Women only: patient must have undergone mammography screening within the last 3 years

Exclusion Criteria:

* older adults with dementia
* older adults with a history of colon cancer
* older adults whose last colonoscopy was read as abnormal
* older women who have a history of breast cancer
* older adults whose PCP has already had 5 patients participate in the study
* older women whose last mammogram was read as abnormal

Ages: 76 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mara A Schonberg, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - BIDMC Affiliated Physicians Group, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schonberg MA, Karamourtopoulos M, Jacobson AR, Aliberti GM, Pinheiro A, Smith AK, Davis RB, Schuttner LC, Hamel MB. A Strategy to Prepare Primary Care Clinicians for Discussing Stopping Cancer Screening With Adults Older Than 75 Years. Innov Aging. 2020 Jul 7;4(4):igaa027. doi: 10.1093/geroni/igaa027. eCollection 2020. PMID 32793815

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prognosis Information and Provider Scripts
Started | 90
Completed | 90
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adults aged 76-89 seen at primary care practices in Boston.
Arm/Group | Prognosis Information and Provider Scripts
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.0 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 79
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Change in Intentions to be Screened for Colorectal Cancer.
Description: Intentions to be screened was measured in a pretest-survey and again within 2 weeks of a PCP visit using the choice/predisposition scale which is measured from 1-15 on a 15 point scale. A score of 1 means that a person does not intend to be screened. A score of 15 means that the person does intend to be screened. A score of 8 means they are unsure. Scores between 2-7 means the person is leaning towards not being screened. A score of 9-14 means that person is leaning towards being screened. We examined the change in intentions to be screened from pretest to the posttest survey. The mean delta was determined at the time of the post-test survey which was completed within two weeks of the PCP visit.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prognosis Information and Provider Scripts
Number analyzed (Participants) | 90
score on a scale | 2.5 (1.9)
Statistical Analysis 1: Comparison: Prognosis Information and Provider Scripts; This was an exploratory and descriptive study to learn if it was feasible to provide PCPs with their patients (aged 76-89) with information about their 10-year prognosis and engage in shared decision making around stopping screening. We measured among the 90 patients that the 45 PCPs saw whether their intentions to be screened declined after seeing their PCP; Test type: Other — Because the observations were matched by the patient, we used the Wilcoxon signed-rank test, a nonparametric paired test; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 2.5 — This was a descriptive feasibility study; This was a descriptive feasibility study
Statistical Analysis 2: Comparison: Prognosis Information and Provider Scripts; This was a descriptive feasibility study; Test type: Other — This was a descriptive feasibility study; p < 0.001, Wilcoxon (Mann-Whitney); Risk Difference (RD) = 0.05; Because the observations were matched by the patient, we used the Wilcoxon signed-rank test, a nonparametric paired test

ADVERSE EVENTS:
Time Frame: 1 week. Patients completed a pre-test survey 3-12 weeks before a PCP visit and then completed a post-test survey immediately after or within 2 weeks of a primary care visit where they may have discussed stopping cancer screening with their PCP.
Arm/Group | Prognosis Information and Provider Scripts
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT03480282/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT03480282/ICF_001.pdf